CLINICAL TRIAL: NCT06289829
Title: Dose Finding Study of Remifentanil for Laryngeal Mask Airway Insertion During Induction Using Remimazolam
Brief Title: The Appropriate Remifentanil Dose for Optimal Insertion of Laryngeal Mask Airway in Adult Patients During Induction of General Anesthesia Using Remimazolam.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 4-2023-1605
Record Dates: First submitted 2024-02-07; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Adult, Laryngeal Masks, Remimazolam, Remifentanil
MeSH Terms: interventions — Airway Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remifentanil (Other): Ambu Auragain inserted after general anesthesia induced with remimazolam and remifentanil
  Interventions: Drug: remifentanil of the assigned dose; Device: Ambu Auragain for airway management

INTERVENTIONS:
Drug: remifentanil of the assigned dose — Ambu Auragain will be inserted after general anesthesia is induced with remimazolam and remifentanil. Each patient will be assigned with a certain dose of remifentanil, according to whether the previous patient's LMA insertion process was successful or not.
Device: Ambu Auragain for airway management — Ambu Auragain, a type of laryngeal mask airway, will be inserted into every patient after general anesthesia has been induced.

SUMMARY:
The laryngeal mask airway (LMA) is an airway maintenance device that is easy to insert and has the advantage of causing less sore throat and autonomic nervous system stimulation. To appropriately insert the LMA, an adequate depth of anesthesia is essential. Various drugs have been studied for inducing anesthesia to achieve the appropriate depth for LMA insertion, and the newly developed benzodiazepine, remimazolam, is gaining attention as one of them. Remimazolam has rapid onset and recovery times, hemodynamic stability, and is often co-administered with opioids like remifentanil for more effective LMA insertion. This study aims to find the optimal dose of remifentanil for the proper insertion of the Ambu Auragain, one of the recently developed LMAs, during induction of anesthesia using remimazolam and the Biased-Coin Up-and-Down method will be used for this purpose. Starting with an initial concentration of remifentanil of 3.0 μg/mL, the success or failure of LMA insertion will determine the dosage for the next subject. Data will be collected from a total of 60 patients, and subsequent analysis will be conducted.

DETAILED DESCRIPTION:
1.Screening Method:

1. Subject screening is conducted based on the results of general preoperative tests, including checking the patient's medical and medication history, routine blood tests, general chemistry and coagulation tests, electrocardiogram (ECG), chest X-ray, etc.
2. Subjects are selected from adult patients undergoing elective surgery under general anesthesia using the LMA within 3 hours.
3. Patients are visited the day before the surgery. Information about the study is provided and patients are allowed sufficient time for deciding participation until arriving at the operating room. Informed consent for the participation is achieved on the morning of surgery.

2.Research Method:

1. Monitoring devices, including electrocardiogram, non-invasive blood pressure monitor, pulse oximeter, and SedLine® brain function monitor (Masimo, Irvine, CA), are applied for patient monitoring according to standard care.
2. Proper insertion of the intravenous catheter in the patient is confirmed. The intravenous line is connected to remifentanil and remimazolam (diluted to concentrations of 20μg/mL and 1mg/mL respectively) using syringe pumps.

(3)100% oxygen is administered at 6L/min for 3 minutes for preoxygenation. (4)Continuous infusion of remifentanil is started using Target-Controlled Infusion (TCI) with the Minto model, adjusting the effect-site concentration based on the biased-coin up-and-down method. The initial concentration for the first patient is 3.0μg/mL. Subsequent doses are determined based on the success or failure of the previous subject's LMA insertion. 0.3mg/kg of remimazolam is simultaneously administered over approximately 10-20 seconds.

(5)100% oxygen is supplied through a facemask and manual ventilation is performed if necessary. When the desired effect-site concentration of remifentanil is confirmed 120 seconds after remimazolam administration, LMA is inserted. The LMA used for the procedure is Ambu®AuraGainTM (Ambu A/S, Ballerup, Denmark). The size of the LMA is selected according to the manufacturer's guide and lubricating jelly is applied on the LMA before the insertion.

(6)If the LMA is determined to obstruct the airway or be malpositioned, it is removedand mask ventilation is reengaged. The effect-site concentration of remifentanil is increased by 0.3μg/mL, and one minute later, the LMA is inserted for the second time using the same procedure. If the insertion proves unsuccessful despite three attempts following the same approach, tracheal intubation is performed.

(7)Data are collected during LMA insertion and maintenance. Continuous infusion of remimazolam and remifentanil is conducted to maintain PSI score in the range of 25-50 during the surgery. Infusion of the anesthetic agents are stopped when the surgery is finished. The LMA is removed after spontaneous breathing is confirmed and the patient is transferred to the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older and less than 65 years
* ASA physical status classification I, II, or III
* Scheduled for elective surgery lasting within 3 hours under general anesthesia using a laryngeal mask

Exclusion Criteria:

* Refusal to participate in the study
* Unable to read the consent form or comprehend the research process (e.g., illiteracy, foreign nationality, cognitive impairment)
* Anatomic structures that are anticipated to cause difficulty in mask ventilation
* History of difficulty in airway management
* Upper respiratory infections or respiratory conditions (e.g., asthma, pneumonia)
* Risk of aspiration (e.g., gastroesophageal reflux)
* Allergies to anesthesia-related drugs, such as benzodiazepines or opioid analgesics
* Impaired liver or kidney function
* Pregnant or breastfeeding patients
* Obesity (body mass index > 30 kg/m2)
* History of drug or alcohol abuse.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-03-02 (Estimated); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Success/failure of LMA insertion on the first attempt | LMA insertion is assessed after inserting the LMA and conducting manual ventilation via the LMA
  LMA insertion is assessed as 'successful' when the following criteria are satisfied.
  * Absence of bucking, laryngospasm, or movements of the head or the limbs during the insertion.
  * Mouth opening is evaluated as 1 or 2 according to the Muzi score. (Muzi score: 1 fully relaxed, 2 mild resistance, 3 tight but opens, 4 closed)
  * Symmetrical chest wall movement and a rectangular capnographic wave is seen when manual ventilation conducted via the inserted LMA.

SECONDARY OUTCOMES:
Difficulty of LMA insertion | Immediately after LMA insertion
  Evaluated as one of 'easy', 'moderate', 'difficult', or 'impossible'.
Optimality of the LMA insertion based on the administered remifentanil dose | Within one minute after LMA insertion
  Evaluated as optimal if swallowing, coughing and gagging, head or body movement, and laryngospasm are absent.
  * 'Swallowing' is evaluated as one of 'absent', 'slight', or 'gross'
  * 'Coughing and gagging' is evaluated as one of 'absent', 'slight', or 'gross'
  * 'Head or body movement' is evaluated as one of 'absent', 'slight', or 'gross'
  * 'Laryngospasm' is evaluated as one of 'absent', 'partial', or 'total'
The number of attempts required for successful LMA insertion and whether intubation was performed. | After a stable airway for the surgery has been achieved.
Air leak volume during positive-pressure ventilation | Tidal volume is set to 8mL/kg immediate after LMA insertion.
  Inspiratory and expiratory volumes are checked to determine air leak volume and peak inspiratory pressure is measured using the anesthesia machine.
Systolic blood pressure | Baseline before induction of anesthesia, immediately before LMA insertion, immediately after successful LMA insertion, 10 minutes after LMA insertion, end of the surgery, 30 minutes after admission to the recovery room
  Baseline before induction of anesthesia, immediately before LMA insertion, immediately after successful LMA insertion, 10 minutes after LMA insertion, end of the surgery, 30 minutes after admission to the recovery room
Heart rate | Baseline before induction of anesthesia, immediately before LMA insertion, immediately after successful LMA insertion, 10 minutes after LMA insertion, end of the surgery, 30 minutes after admission to the recovery room
Patient State Index (PSI) | Baseline before induction of anesthesia, immediately before LMA insertion, immediately after successful LMA insertion, 10 minutes after LMA insertion, End of the surgery, 30 minutes after admission to the recovery room
Severity of hoarseness | 30 minutes after admission to the recovery room Outcome measure assemssent - Evaluated as one of 'none', 'mild', 'moderate', or 'severe'
Severity of coughing | 30 minutes after admission to the recovery room Outcome measure assemssent - Evaluated as one of 'none', 'less than a common cold', 'similar to a common cold', or 'more than a common cold'
Severity of sore throat | 30 minutes after admission to the recovery room Outcome measure assemssent - Evaluated as one of 'none', 'less than a common cold', 'similar to a common cold', or 'more than a common cold'
Diastolic blood pressure | Baseline before induction of anesthesia, immediately before LMA insertion, immediately after successful LMA insertion, 10 minutes after LMA insertion, end of the surgery, 30 minutes after admission to the recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No